CLINICAL TRIAL: NCT01905995
Title: Recording of Gait and Speech Related Neurophysiological Parameters With an Implantable Bi-directional Deep Brain Stimulation System in Parkinson's Disease
Brief Title: Basal Ganglia Local Field Potentials in Gait and Speech
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kai Bötzel (Other)
Collaborators: Medtronic (Industry); Lueneburg Heritage (Unknown)
Responsible Party: Sponsor-Investigator, Kai Bötzel, Professor Dr. med., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: BG EEG Munich
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Basal Ganglia Diseases
Keywords: deep brain sitimulation; local field potentials
MeSH Terms: conditions — Basal Ganglia Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced Parkinson's disease: no intervention - observational study

SUMMARY:
Electrid activity of the basal ganglia will be recorded with an implantable deep brain stimulation device (supplied by Medtronic Inc).

Study hypothesis is that these activities differ according to what the patient does, i.e. are different during gait and speech.

ELIGIBILITY:
Inclusion Criteria:

* good levodopa response

Exclusion Criteria:

* dementia

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Difference of frequency spectrum of basal ganglia local field potentials during gait and speech | 1 year

SECONDARY OUTCOMES:
Evidence for the benefit of different stimulator settings for gait and speech | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kai Bötzel, M.D., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Dept. of Neurology, Ludwig-Maximilians University of Munich, Munich/München, Germany